CLINICAL TRIAL: NCT07305090
Title: Development of a Multi-biomarker Panel for Prognostic Stratification and Treatment Response Prediction in Acute Graft Versus Host Disease of the Gut
Acronym: GUT-PREDICTION
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: GUT-PREDICTION; RC-2025-2794670 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2025-11-24; First posted 2025-12-26 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Blood Cancer
Keywords: GvHD; aGvHD; GI
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, saliva, stool, urine, bowel biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hematological diseases treated with allogeneic hematopoietic cell transplantation
  Interventions: Other: Adult and pediatric patients with hematological diseases treated with allogeneic hematopoietic cell transplantation

INTERVENTIONS:
Other: Adult and pediatric patients with hematological diseases treated with allogeneic hematopoietic cell transplantation — The specific activities planned for the study will be:
  * collection of blood, saliva, stool, and urine samples
  * during colonoscopy or esophagogastroduodenoscopy, two biopsies will be taken for molecular biology analysis
  * administration of a food diary together with a questionnaire on eating habits, to be completed by the patient on the days of scheduled visits during the course of therapy, in conjunction with the collection of stool samples.
  * assessment of in vivo permeability using sugar tests.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is a life-saving treatment for many malignant hematologic diseases. Its curative potential is due to both high-dose chemotherapy and the graft-versus-host disease (GvHD) process, in which the donor's T cells recognize the recipient's tissue as foreign. However, GvHD is a potentially fatal complication that significantly affects both survival and quality of life. GvHD can be acute or chronic, and one of the main target organs involved in acute GvHD is the intestine, with a high rate of treatment failure and mortality. We expect to identify a set of biomarkers, both clinical and experimental, that will enable the stratification of patients based on prognosis and response to treatment in intestinal GvHD. The ultimate goal of the study is to integrate clinical, transplant, and biomarker data into a robust predictive algorithm. This tool will enable personalized therapeutic approaches based on early biomarkers, improving prognostic accuracy for patient outcomes and optimizing therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 12 years
* Indication for allogeneic HSCT
* Obtaining informed consent

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be constituted through the consecutive enrollment of adult and pediatric patients with hematological diseases treated with allogeneic hematopoietic cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Identify a set of biomarkers capable of stratifying the overall risk of developing grade 2-4 GI GVHD in adult and pediatric patients with hematological diseases undergoing allogeneic hematopoietic cell transplantation. | Between the infusion of the transplant and the following 120 days

SECONDARY OUTCOMES:
Identification of biomarkers for mortality risk stratification and immunological and nutritional profiling in GvHD | After the start of therapy. Nutritional aspects will be assessed upon the patient's admission to the ward and at the onset of the event (GVHD)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No